CLINICAL TRIAL: NCT02409719
Title: Home Rehabilitation in Patients After Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, FELIX VILCHEZ CAVAZOS, MD-PhD, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR14-005
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis; Rehabilitation
Keywords: Arthritis, Degenerative; Recovery of function
MeSH Terms: conditions — Osteoarthritis | interventions — Appointments and Schedules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control - Verbal information and Booklet (Active Comparator): Verbal information will be provided in order to explain how the patient should perform physical rehabilitation exercises. Furthermore, an illustrative booklet with representative exercises will be given.
  Interventions: Other: Verbal Information and Booklet
- Study - Verbal information, Booklet & Schedule. (Experimental): Verbal information will be provided in order to explain how the patient should perform physical rehabilitation exercises. Furthermore, an illustrative booklet with representative exercises will be given. Also, an illustrative daily schedule to mark on the exact day in which the exercise was performed
  Interventions: Other: Schedule; Other: Verbal Information and Booklet

INTERVENTIONS:
Other: Schedule — Illustrative daily planner to point the day that the exercise was performed
  Other Names: Planner
  Arms: Study - Verbal information, Booklet & Schedule.
Other: Verbal Information and Booklet — Verbal information will be provided in order to explain how the patient should perform physical rehabilitation exercises. Furthermore, an illustrative booklet with representative exercises will be given. Also, an illustrative daily schedule to mark on the exact day in which the exercise was performed
  Other Names: Verbal and Booklet Physical Rehabilitation information

SUMMARY:
The investigators include patients attending the outpatient clinic in the area of Orthopedics and Traumatology of the investigators hospital with a diagnosis of knee osteoarthritis, which treatment requires surgery. Patients will be divided into two groups. In both groups, they will be given verbal, clear and detailed information on the approach to follow, the exercises given in brochures, and in the study group a schedule will be given in order to record rehabilitation exercises in patients after total knee replacement (TKA). Both groups will be assessed before and after surgery, together with outpatient follow-up by, WOMAC, Visual Analogue Scale and OKS (Oxford Knee Score).

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common rheumatic disease worldwide. OA cause joint pain and occupational disability in the adult population. In Mexico, OA is one of the top ten reasons of consultation in primary attention care.

Joint arthroplasty is a major advance in the treatment of chronic joint pain. It is indicated in patients in whose conservative medical therapy has failed. Total knee arthroplasty (TKA) is a surgery that reduces pain and improves function and quality of life in patients with knee disorders, actually is one of the most successful medical procedures. However, a critical consideration in patients with TKA is the successful control of postoperative pain. An adequate pain control allows faster rehabilitation, reduces complications and is highly correlated with patient satisfaction. A multimodal pain management decreases the use of narcotics, improve pain scores, increase patient satisfaction and allows early recovery.

Regarding postoperative rehabilitation, its suggested that rehabilitation programs are based on a biopsychosocial philosophy and integrate exercises and self-management interventions are effective in the treatment of osteoarthritis. Rehabilitation therapy an important area that should be considered. It helps people recover faster from their illness, injury or medical procedures and make possible to get back to their daily activities.

The World Health Organization describes rehabilitation as a process that aims to enable people to maintain and achieve their physical, sensory, intellectual, functional, psychological and social level in an optimal way. It is known that rehabilitation involves contributions from various health disciplines, including physical therapy and occupational therapy and offered in inpatient, outpatient and community patients.

In patients with total knee replacement, rehabilitation interventions may involve education and exercise before surgery, early mobilization while being in the hospital and a postoperative program, along with an adequate pain management.

Perioperative care has shown an improvement in the recovery, it reduces hospital day stay, convalescent and risk of postoperative medical complications.

It has been shown that early initiation of rehabilitation within 24 hours after total knee arthroplasty reduces in-hospital time and decreases the number of sessions required to achieve autonomy, balance and normal gait. Madsen et al. demonstrated that rehabilitation exercises at home have the same effect as those made in rehabilitation group within six months postoperatively, based on a study of 80 patients randomly divided into a control- study group.

Optimal pain management is vital seeking to achieve the goal of recovery called fast track. It involves early therapy with specialized protocols, early discharge and quick recovery. Lamplot et al. demonstrated in a prospective randomized study of 36 patients, using this method, a decrease in opioid consumption and its adverse effects, a decreased pain score, a shortening time for physical therapy and an increase in patient satisfaction.

Postoperative analgesia can be achieved by a variety of techniques. These include: intravenous analgesia, epidural analgesia, techniques for peripheral nerve block and periarticular injections. All aim to control pain in patients and provide the better satisfaction.

Integrating these interventions in a clinical pathway, better functional results are obtained, hospital stay is reduced and there is an improvement in the patient's recovery, mainly in short-term.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years
* Patients with Knee osteoarthritis (OA) grade 4 ( Kellgren-Lawrence based on radiographic findings)
* Total Knee Arthroplasty (TKA) for primary OA
* Rapid rehabilitation desire

Exclusion Criteria:

* Age <18 and > 90 years
* Patients with Knee osteoarthritis grade 1-2 ( Kellgren-Lawrence based on radiographic findings)
* Patients with asociated Rheumatic syndromes
* Patients with anticoagulant therapy
* Patients with hepatic problems, Diabetes Mellitus, Coagulopathy, hearth conditions, immunodepressed, or infections
* Drugs abuse history
* Physiatric disease
* Pregnant patients
* Patients with hemoglobin values < 11g/dl , platelets < 150,000/ μL

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-07; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Vilchez, MD-PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Facultad de Medicina UANL, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Minns Lowe CJ, Barker KL, Dewey M, Sackley CM. Effectiveness of physiotherapy exercise after knee arthroplasty for osteoarthritis: systematic review and meta-analysis of randomised controlled trials. BMJ. 2007 Oct 20;335(7624):812. doi: 10.1136/bmj.39311.460093.BE. Epub 2007 Sep 20. PMID 17884861
- [Background] Meier W, Mizner RL, Marcus RL, Dibble LE, Peters C, Lastayo PC. Total knee arthroplasty: muscle impairments, functional limitations, and recommended rehabilitation approaches. J Orthop Sports Phys Ther. 2008 May;38(5):246-56. doi: 10.2519/jospt.2008.2715. Epub 2007 Dec 14. PMID 18448878
- [Background] Labraca NS, Castro-Sanchez AM, Mataran-Penarrocha GA, Arroyo-Morales M, Sanchez-Joya Mdel M, Moreno-Lorenzo C. Benefits of starting rehabilitation within 24 hours of primary total knee arthroplasty: randomized clinical trial. Clin Rehabil. 2011 Jun;25(6):557-66. doi: 10.1177/0269215510393759. Epub 2011 Mar 7. PMID 21382863
- [Background] Kauppila AM, Sintonen H, Aronen P, Ohtonen P, Kyllonen E, Arokoski JP. Economic evaluation of multidisciplinary rehabilitation after primary total knee arthroplasty based on a randomized controlled trial. Arthritis Care Res (Hoboken). 2011 Mar;63(3):335-41. doi: 10.1002/acr.20398. Epub 2010 Nov 15. PMID 21080347
- [Background] DiSotto-Monastero M, Chen X, Fisch S, Donaghy S, Gomez M. Efficacy of 7 days per week inpatient admissions and rehabilitation therapy. Arch Phys Med Rehabil. 2012 Dec;93(12):2165-9. doi: 10.1016/j.apmr.2012.07.003. Epub 2012 Jul 20. PMID 22819810
- [Background] Ribinik P, Le Moine F, de Korvin G, Coudeyre E, Genty M, Rannou F, Yelnik A, Calmels P. Physical and rehabilitation medicine (PRM) care pathways: "patients after total knee arthroplasty". Ann Phys Rehabil Med. 2012 Nov;55(8):533-9. doi: 10.1016/j.rehab.2012.02.001. Epub 2012 Mar 3. PMID 22455993
- [Background] Bandholm T, Kehlet H. Physiotherapy exercise after fast-track total hip and knee arthroplasty: time for reconsideration? Arch Phys Med Rehabil. 2012 Jul;93(7):1292-4. doi: 10.1016/j.apmr.2012.02.014. Epub 2012 Feb 27. PMID 22494947
- [Background] Nakai T, Tamaki M, Nakamura T, Nakai T, Onishi A, Hashimoto K. Controlling pain after total knee arthroplasty using a multimodal protocol with local periarticular injections. J Orthop. 2013 Mar 17;10(2):92-4. doi: 10.1016/j.jor.2013.02.001. eCollection 2013. PMID 24403757
- [Background] Madsen M, Larsen K, Madsen IK, Soe H, Hansen TB. Late group-based rehabilitation has no advantages compared with supervised home-exercises after total knee arthroplasty. Dan Med J. 2013 Apr;60(4):A4607. PMID 23651717
- [Background] Ibrahim MS, Khan MA, Nizam I, Haddad FS. Peri-operative interventions producing better functional outcomes and enhanced recovery following total hip and knee arthroplasty: an evidence-based review. BMC Med. 2013 Feb 13;11:37. doi: 10.1186/1741-7015-11-37. PMID 23406499
- [Background] Lamplot JD, Wagner ER, Manning DW. Multimodal pain management in total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Feb;29(2):329-34. doi: 10.1016/j.arth.2013.06.005. Epub 2013 Jul 11. PMID 23850410
- See also: Epidemiology of Knee and Hip Arthroplasty: A Systematic Review — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3092498/
- See also: Total Joint Replacement Rehabilitation — http://emedicine.medscape.com/article/320061-overview

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was held in the outpatient clinic in the area of Orthopedics and Traumatology of the investigators hospital with a diagnosis of knee osteoarthritis, which treatment requires surgery in which the recruitment process started June 2014 until January 2019.
  The objective was to recruit 76 patients were randomly divided into two groups.
Pre-assignment Details: 6 patients were lost to follow up.
Groups:
- Control - Verbal Information and Booklet: Verbal information will be provided in order to explain how the patient should perform physical rehabilitation exercises. Furthermore, an illustrative booklet with representative exercises will be given.
  Verbal Information and Booklet: Verbal information will be provided in order to explain how the patient should perform physical rehabilitation exercises. Furthermore, an illustrative booklet with representative exercises will be given. Also, an illustrative daily schedule to mark on the
- Study - Verbal Information, Booklet & Schedule.: Verbal information will be provided in order to explain how the patient should perform physical rehabilitation exercises. Furthermore, an illustrative booklet with representative exercises will be given. Also, an illustrative daily schedule to mark on the exact day in which the exercise was performed
  Schedule: Illustrative daily planner to point the day that the exercise was performed
  Verbal Information and Booklet: Verbal information will be provided in order to explain how the patient should perform physical rehabilitation exercises. Furthermore, an illustrative booklet with representative exercises will be given. Also, an illustrative daily schedule to mark on the
Period: Overall Study
Arm/Group | Control - Verbal Information and Booklet | Study - Verbal Information, Booklet & Schedule.
Started (Each milestone corresponds to the time of evaluation.) | 31 | 45
2 Weeks | 28 | 42
4 Weeks | 28 | 42
6 Weeks | 28 | 42
3 Months | 28 | 42
6 Months | 28 | 42
12 Months | 28 | 42
Completed | 28 | 42
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Verbal Information and Booklet | Study - Verbal Information, Booklet & Schedule. | Total
Number analyzed (Participants) | 28 | 42 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 14 | 22
  >=65 years | 20 | 28 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 22 | 34
  Male | 16 | 20 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Knee right or left [Number; unit: participants]
  Right Knee | 14 | 24 | 38
  Left Knee | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Total WOMAC Score
Description: The total score is provided for Western Ontario and McMaster Universities Arthritis Index (WOMAC).
  It is a widely score used in the evaluation of Hip and Knee Osteoarthritis. Consists of a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  pain (5 items), stiffness (2 items), and physical functioning (17 items) of the joints.
  * Scale Range: 5 items of pain (score range 0-20), 2 items for stiffness (score range 0-8), and 17 items for functional limitation (score range 0-68). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Total WOMAC score range 0-96.
  * For each subscale higher values represent worse outcomes.
  * Subscales are summed for a total WOMAC score. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
  WOMAC Index was developed in 1982 at Western Ontario and McMaster Universities.
Time Frame: up to 12 months (O, 2, 4, 6 weeks, 3,6 and 12 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Verbal Information and Booklet | Study - Verbal Information, Booklet & Schedule.
Number analyzed (Participants) | 28 | 42
score on a scale
  0 weeks | 51.64285714 (17.26957137) | 52.47619048 (20.96947619)
  2 weeks | 39.60714286 (18.01920639) | 40.38095238 (16.73458866)
  4 weeks | 29.42857143 (13.48916869) | 30.85714286 (14.35197178)
  6 weeks | 25.32142857 (16.60444735) | 24.88095238 (14.11140756)
  3 months | 16 (11.18861856) | 20.19047619 (11.89842805)
  6 months | 10.28571429 (7.721337165) | 14.11904762 (8.969330891)
  12 months | 6.571428571 (6.941173833) | 9.166666667 (7.525296094)

2. Secondary Outcome: Visual Analog Scale (Measure of Pain Intensity)
Description: The pain Visual Analog Scale is a unidimensional measure of pain intensity. The scale is most commonly anchored by "no pain " (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (scale of 10).
Time Frame: up to 12 months (O, 2, 4, 6 weeks, 3,6 and 12 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Verbal Information and Booklet | Study - Verbal Information, Booklet & Schedule.
Number analyzed (Participants) | 28 | 42
score on a scale
  0 weeks | 8.178571429 (1.906199854) | 8.285714286 (1.8251056)
  2 weeks | 5.392857143 (2.114137346) | 5.714285714 (2.051599189)
  4 weeks | 4 (1.943650632) | 4.261904762 (2.012879551)
  6 weeks | 3 (2.388242807) | 3.333333333 (2.385593618)
  3 months | 2.214285714 (2.266619981) | 2.619047619 (2.197031045)
  6 months | 1.428571429 (1.687175405) | 1.785714286 (1.746574547)
  12 months | 0.678571429 (0.944911183) | 0.761904762 (1.225929688)

3. Other Pre Specified Outcome: Oxford Knee Score (OKS)
Description: The Oxford Knee Score is a 12-item patient-reported outcome specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty). It is short, reproducible, valid and sensitive to clinically important changes.
  Consists of 12 multiple choice questions consisting of five answers with a maximum score of 60.
  Score ranges
  * Score 0 to 19: May indicate severe knee arthritis. It is highly likely that you may well require some form of surgical intervention, contact your family physician for a consult with an Orthopaedic Surgeon.
  * Score 20 to 29: May indicate moderate to severe knee arthritis. See your family physician for an assessment and x-ray. Consider a consult with an Orthopaedic Surgeon.
  * Score 30 to 39: May indicate mild to moderate knee arthritis. Consider seeing your family physician for an assessment and possible x-ray. You may benefit from non-surgical treatment, such as exercise, weight loss, and /or anti-inflammatory med
Time Frame: up to 12 months (O, 2, 4, 6 weeks, 3,6 and 12 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control - Verbal Information and Booklet | Study - Verbal Information, Booklet & Schedule.
Number analyzed (Participants) | 28 | 42
units on a scale
  0 weeks | 17.10714286 (6.436811298) | 17.45238095 (8.554566263)
  2 weeks | 22.60714286 (7.568645291) | 21.35714286 (7.367765749)
  4 weeks | 28.5 (5.666666667) | 25.90243902 (7.059762312)
  6 weeks | 32 (7.693190832) | 30.02380952 (7.202601479)
  3 months | 36.89285714 (6.020577588) | 33.54761905 (6.868813868)
  6 months | 38.78571429 (7.067699835) | 37.42857143 (5.926965485)
  12 months | 41.21428571 (5.902649392) | 40.54761905 (4.357233296)

ADVERSE EVENTS:
Time Frame: up to 12 months
Arm/Group | Control - Verbal Information and Booklet | Study - Verbal Information, Booklet & Schedule.
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/42
Other Adverse Events (participants affected / at risk) | 0/28 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control - Verbal Information and Booklet (N=28) | Study - Verbal Information, Booklet & Schedule. (N=42)
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Required Hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT02409719/Prot_SAP_000.pdf